CLINICAL TRIAL: NCT05460793
Title: Dutch ICH Surgery Trial; Minimally Invasive Endoscopy-guided Surgery for Spontaneous Supratentorial Intracerebral Hemorrhage
Brief Title: Dutch Intracerebral Hemorrhage Surgery Trial
Acronym: DIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch National Health Care Institute (Other); Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL80112.078.22
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Intracerebral Hemorrhage; Minimally Invasive Surgical Procedures; Endoscopic Surgical Procedures
Keywords: Intracerebral Hemorrhage; Surgical Procedures, Minimally Invasive; Surgical Procedures, Endoscopic
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: prospective, randomized, open, blinded endpoint (PROBE) clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Surgical treatment (Experimental): Minimally invasive endoscopy-guided surgery in addition to standard medical management for the treatment of spontaneous supratentorial intracerebral hemorrhage performed within 8 hours of symptom onset.
  Interventions: Device: Minimally invasive endoscopy-guided surgery
- Standard medical management (No Intervention): Standard medical treatment for the treatment of spontaneous supratentorial intracerebral hemorrhage (treatment of blood pressure, admission to stroke unit and supportive care, surgical treatment if necessary in case of deterioration).

INTERVENTIONS:
Device: Minimally invasive endoscopy-guided surgery — The devices allowed into the trial, are minimally invasive neuronavigation integrated endoscopy-guided devices that are CE approved and admissible by the steering committee. Currently, only the Artemis Neuro Evacuation Device (Penumbra Inc, Alameda, California, USA) is available and CE approved.
  Arms: Surgical treatment

SUMMARY:
Background: Intracerebral hemorrhage (ICH) accounts for 16-19% of all strokes in Western Europe and contributes profoundly to mortality and disability. Thirty-day case fatality is 40% and of those surviving, only few gain independence. Except for stroke unit care and possibly early blood pressure lowering, there is currently no treatment of proven benefit. Surgical treatment has so far not been proven effective. In the largest trials STICH I and II, and MISTIE III, the median time to treatment was more than 24 hours, which may be an important explanation for the lack of a treatment effect. A recent meta-analysis of randomized controlled trials showed that surgical treatment may be beneficial, in particular with minimally invasive procedures and when performed early. In the Dutch ICH Surgery pilot study, we showed that early minimally invasive endoscopy-guided surgical treatment performed within 8 hours of symptom onset in patients with supratentorial ICH is safe and technically effective. We hypothesize that early minimally invasive endoscopy-guided surgery improves the outcome in patients with supratentorial spontaneous ICH.

Objectives:

1. To study whether minimally invasive endoscopy-guided surgery, in addition to standard medical management, for the treatment of spontaneous supratentorial ICH performed within 8 hours of symptom onset, improves functional outcome in comparison with standard medical management alone;
2. Determine whether patients treated with minimally invasive surgery develop less perihematomal edema on non-contrast CT at day 6 (±1 day) than controls, and whether the CT perfusion permeability surface-area product around the ICH at baseline modifies this effect (DIST-INFLAME);
3. Compare immune profiles over time in peripheral venous blood between surgically treated patients and controls (DIST-INFLAME);
4. To assess the cost-effectiveness and budget-impact of minimally invasive endoscopy-guided surgery for the treatment of spontaneous supratentorial ICH performed within 8 hours of symptom onset.

Study design: A multicenter, prospective, randomized, open, blinded endpoint clinical trial.

Study population: We aim to include 600 patients of ≥ 18 years with a spontaneous supratentorial ICH with a hematoma volume of ≥ 10 mL and a NIHSS of ≥ 2. Patients with an aneurysm, arteriovenous malformation (AVM), dural arteriovenous fistula (DAVF), or cerebral venous sinus thrombosis (CVST) as cause of their ICH will be excluded based on the admission CT-angiography. Patients with a known tumor or cavernoma will also be excluded. For DIST-INFLAME (the second and third objective), we will include 200 patients; 100 randomized to intervention and 100 randomized to standard medical management.

Intervention: Patients will be randomized (1:1) to minimally invasive endoscopy-guided surgery performed within 8 hours of symptom onset in addition to standard medical management or to standard medical management alone.

Primary study outcome: the modified Rankin scale (mRS) score at 180 days. The treatment effect will be estimated with ordinal logistic regression analysis as common odds ratio, adjusted for prespecified prognostic factors.

Secondary outcomes: mRS score at 90 and 365 days; favorable outcome (defined as a mRS 0-2 and 0-3) and all other possible dichotomizations of the mRS at 90, 180 and 365 days; NIHSS at day 6 (±1 day); death, Barthel Index, EuroQol-5D-5L, SS-QOL, iMCQ, iPCQ and iVICQ at 90, 180 and 365 days. Safety outcomes will be death within 24 hours, at 7 and at 30 days and procedure-related complications within 7 days. Technical effectiveness outcomes will be percentage volume reduction based on the baseline CT and CT at 24 hours (± 6 hours), percentage of participants with clot volume reduction ≥70%, and ≥80%, and with remaining clot volume ≤10mL, and ≤15mL, and conversion to craniotomy. In DIST-INFLAME, outcomes will include perihematomal edema at 6 days (±1 day), functional outcome at 180 days and immune and metabolomic profiles at 3 (± 12 hours) and 6 days (±1 day).

DETAILED DESCRIPTION:
The full protocol is available at: http://dutch-ich.nl/

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. NIHSS ≥ 2;
3. Supratentorial non-traumatic ICH confirmed by non-contrast CT, without a CT-angiography confirmed causative vascular lesion (e.g. aneurysm, arteriovenous malformation [AVM], dural arteriovenous fistula [DAVF], cerebral venous sinus thrombosis [CVST]), or other known underlying lesion (e.g. tumor, cavernoma);
4. Minimal hematoma volume of 10 mL;
5. Intervention can be started within 8 hours of symptom onset;
6. Written informed consent (deferred).

Exclusion Criteria:

1. Considerable pre-stroke dependency in activities of daily living, defined as a pre-stroke mRS ≥3;
2. ICH-GS score ≥11;
3. Hemorrhage due to hemorrhagic transformation of an infarct;
4. Untreated coagulation abnormalities, including INR >1.3 (point of care measurement allowed), treatment with heparin and treatment with factor Xa inhibitors. Patients on vitamin K antagonist can be included after correction of the INR, and patients on dabigatran (direct thrombin inhibitor) can be included after reversal of dabigatran with idarucizumab;
5. Moribund (e.g. coning, bilateral dilated unresponsive pupils), or progressively deteriorating clinical course with imminent death;
6. Pregnancy (note: most patients will be beyond childbearing age);
7. DIST-INFLAME sub-study: patients that use immunosuppressive or immune-modulating medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) at 180 days | 180 days (±14 days)
  Ordinal shift in functional outcome assessed with the mRS at 180 days, adjusted for prespecified prognostic factors. This is a six point scale in which a score of 0 means no symptoms at all, a higher score means more impairment, and a score of 6 means the participant is dead.

SECONDARY OUTCOMES:
mRS at 90 days | 90 days (±14 days)
mRS at 365 days | 365 days (±14 days)
Favorable outcome, defined as a mRS of 0-2 at 90 days | 90 days (±14 days)
Favorable outcome, defined as a mRS of 0-2 at 180 days | 180 days (±14 days)
Favorable outcome, defined as a mRS of 0-2 at 365 days | 365 days (±14 days)
Favorable outcome, defined as a mRS of 0-3 at 90 days | 90 days (±14 days)
Favorable outcome, defined as a mRS of 0-3 at 180 days | 180 days (±14 days)
Favorable outcome, defined as a mRS of 0-3 at 365 days | 365 days (±14 days)
All other possible dichotomizations of the mRS at 90 days | 90 days (±14 days)
All other possible dichotomizations of the mRS at 180 days | 180 days (±14 days)
All other possible dichotomizations of the mRS at 365 days | 365 days (±14 days)
National Institute of Health Stroke Scale (NIHSS) at 6 days (±1 day) | 6 days (±1 day)
Death at 90 days | 90 days (±14 days)
Death at 180 days | 180 days (±14 days)
Death at 365 days | 365 days (±14 days)
Barthel Index at 90 days | 90 days (±14 days)
Barthel Index at 180 days | 180 days (±14 days)
Barthel Index at 365 days | 365 days (±14 days)
EuroQol 5D-5L at 90 days | 90 days (±14 days)
EuroQol 5D-5L at 365 days | 180 days (±14 days)
EuroQol 5D-5L at 365 days | 365 days (±14 days)
Stroke-Specific Quality of Life scale at 90 days | 90 days (±14 days)
Stroke-Specific Quality of Life scale at 180 days | 180 days (±14 days)
Stroke-Specific Quality of Life scale at 365 days | 365 days (±14 days)
iMTA Medical Consumption Questionnaire (iMCQ) at 90 days | 90 days (±14 days)
iMTA Medical Consumption Questionnaire (iMCQ) at 180 days | 180 days (±14 days)
iMTA Medical Consumption Questionnaire (iMCQ) at 365 days | 365 days (±14 days)
iMTA Productivity Cost Questionnaire (iPCQ) at 90 days | 90 days (±14 days)
iMTA Productivity Cost Questionnaire (iPCQ) at 180 days | 180 days (6 months)
iMTA Productivity Cost Questionnaire (iPCQ) at 365 days | 365 days (±14 days)
iMTA Valuation of Informal Care Questionnaire (iVICQ) at 90 days | 90 days (±14 days)
iMTA Valuation of Informal Care Questionnaire (iVICQ) at 180 days | 180 days (±14 days)
iMTA Valuation of Informal Care Questionnaire (iVICQ) at 365 days | 365 days (±14 days)
Home time at 90 days | 90 days (±14 days)
Home time at 180 days | 180 days (±14 days)
Home time at 365 days | 365 days (±14 days)
Patient location at 90 days | 90 days (±14 days)
Patient location at 180 days | 180 days (±14 days)
Patient location at 365 days | 365 days (±14 days)
Death within 24 hours | 24 hours
Procedure related complications within 7 days | 7 days
Case-fatality at 7 days | 7 days
Case-fatality at 30 days | 30 days
Percentage volume reduction based at 24 hours | 24 hours
  The percentage of volume reduction based on baseline CT and CT at 24 hours (in the intervention group)
Percentage of participants with hematoma volume reduction ≥70% | 24 hours
  The percentage of participants in which the hematoma volume is reduced with 70% or more, based on the baseline CT and CT at 24 hours (in the intervention group)
Percentage of participants with hematoma volume reduction ≥80% | 24 hours
  The percentage of participants in which the hematoma volume is reduced with 80% or more, based on the baseline CT and CT at 24 hours (in the intervention group)
Percentage of participants with remaining hematoma volume ≤10mL | 24 hours
  The percentage of participants in which the hematoma volume is reduced to 10 mL or less, based on the baseline CT and CT at 24 hours (in the intervention group)
Percentage of participants with remaining hematoma volume ≤15mL | 24 hours
  The percentage of participants in which the hematoma volume is reduced to 15 mL or less, based on the baseline CT and CT at 24 hours (in the intervention group)
Conversion to craniotomy | 24 hours
  The percentage of participants in which a conversion to craniotomy was required and done (in the intervention group)

OTHER OUTCOMES:
Perihematomal edema at 6 days (±1 day) | 6 days (±1 day)
  DIST-INFLAME sub-study: Perihematomal edema assessed on non-contrast CT at 6 days (±1 day)
Immune and metabolomic profiles in venous blood at 3 days | 3 days
  DIST-INFLAME sub-study: Immune and metabolomic profiles in venous blood at 3 days
Immune and metabolomic profiles in venous blood at 6 days (±1 day) | 6 days (±1 day)
  DIST-INFLAME sub-study: Immune and metabolomic profiles in venous blood at 6 days (±1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Catharina JM Klijn, MD PhD, Principal Investigator — Radboud University Medical Center; Ruben Dammers, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (11):
- Netherlands (11):
  - Amsterdam University Medical Center, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - Haaglanden Medical Center, The Hague
  - Elisabeth-TweeSteden Hospital, Tilburg
  - University Medical Center Utrecht, Utrecht
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other parties to maximize the usefulness of the collected research data. Data can be requested from the principal investigators with a detailed description of the objectives and methods of the study for which the data is intended. Data will be made available for this purpose at least 18 months after the publication of the main report. Data may also be shared with non-commercial parties for scientific purposes, including individual patient meta-analyses, and with the commercial parties involved in this study as manufacturers of minimally invasive neuronavigation integrated endoscopy-guided devices. For these purposes, specific consent will be asked from the participants. In addition, specific consent will be asked for sharing of de-identified data outside of the European Union.
Time Frame: at least 18 months after the publication of the main report.
Access Criteria: Written proposals will be assessed by DIST investigators for appropriateness of use, and a data sharing agreement in accordance with Dutch regulations will be put in place before data is shared.

REFERENCES:
- [Derived] Wilting FNH, Wolsink A, Colmer NHC, Schreuder FHBM, Brouwers HB, Boogaarts HD, Dippel DWJ, Hannink G, Jolink WMT, Verbaan D, Wermer MJH, Dammers R, Klijn CJM. The Dutch Intracerebral Haemorrhage Surgery Trial: study protocol for a randomised clinical trial of minimally invasive endoscopy-guided surgery in patients with spontaneous, supratentorial intracerebral haemorrhage. Eur Stroke J. 2026 Jan 1;11(1):aakaf008. doi: 10.1093/esj/aakaf008. PMID 41614502
- See also: Website of the Dutch ICH Surgery Trial (DIST) — http://dutch-ich.nl